CLINICAL TRIAL: NCT06804785
Title: Hybrid Intelligence for Trustable Diagnosis and Patient Management of Prostate Cancer (HIT-PIRADS)
Acronym: HIT-PIRADS
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: STU00218692; 5U01CA268808-02 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2025-02-03 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Elevated PSA; Elevated Prostate-Specific Antigen; Abnormal digital rectal exam; Prostate Cancer; Prostate; AI; Artificial Intelligence; Oncology
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Biopsy naïve participants with elevated PSA (4.0-10.0 ng/ml) or abnormal digital rectal exam with PSA of 2.00-10.00 ng/ml as indicated in their lab report.

SUMMARY:
The purpose of this study is to develop a new way to diagnose prostate cancer through the use of artificial intelligence. The goal is for this new method to reduce delays in diagnoses and to avoid invasive procedures such as biopsies.

DETAILED DESCRIPTION:
The overall goal of this project is to create a diagnosis and patient management strategy (called HIT-PIRADS) for prostate cancer (PCa) that will significantly increase positive predictive value (PPV) for clinically significant PCa detection while minimizing unnecessary prostate biopsies and related morbidities. Due to its interpretable nature and bias correction paradigm, the AI system will generate predictions that physicians can trust. One of the immediate outcomes of the system will be a reproducible risk scoring system that can be used in community hospitals and locales without MRI-subspeciality genitourinary trained radiologists to improve the accuracy of prostate imaging nationwide. In the long term, the investigators expect HIT-PIRADS to be widely adopted in clinics and trigger other treatment and prevention strategies to be developed based on HIT-PIRADS.

ELIGIBILITY:
Inclusion Criteria:

* Elevated PSA (4.0-10.0 ng/ml) or abnormal digital rectal exam with PSA of 2.00-10.00 ng/ml as indicated in the patient's lab report.
* Patients must be biopsy naïve, confirmed with patient or medical record.
* Patients must be male, ≥18 and ≤ 89 years of age.
* Patient must have a life expectancy ≥10 years, determined by PI.
* Patients must exhibit an ECOG performance status of 0-2, as noted in their medical record.

Exclusion Criteria:

* Patients who are on a 5-α-reductase inhibitor within 12 months of enrollment, as confirmed by medical record.
* Patients who have had a prostate infection within 1 month of enrollment, as confirmed by medical record.
* Patients who are receiving or who received prostate cancer treatment (e.g., androgen deprivation therapy, surgery, radiation therapy or adjuvant/neoadjuvant therapy with investigational drugs) per their medical record.
* Patients who've had an invasive urological procedure within 1 month of enrollment, as confirmed by their medical record and patient reporting.
* Patients with no access to the rectum for a transrectal ultrasound, as determined by the Urologist.
* Patients with a contraindication to magnetic resonance imaging (MRI).
* Vulnerable populations: Prisoners or adult men >89 years old.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at an increased risk of having prostate cancer. An increased risk for prostate cancer means the patient may have had either a blood test which indicated they have an elevated prostate-specific antigen (PSA) (a protein produced by both cancerous and noncancerous tissue in the prostate), or an abnormal exam of the patient's rectum, anus or prostate gland.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with detection of clinically significant prostate cancer (csPCa) | 01/01/2016-12/31/2026
  csPCa is defined as PCa with a Gleason Grade Group of 2 through 5 found on prostate biopsy. Detection of csPCa will be compared for HITPIRADS vs. PIRADS v2.1 with a focus on suspicious lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes